CLINICAL TRIAL: NCT00004348
Title: Study of Protein Translocation in Patients With Beta-Oxidation Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 199/11907; WUSM-880075R (Other: Washington University School of Medicine); R37DK020407 (NIH)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Beta-Oxidation Disorder; Peroxisomal Disorders
Keywords: beta-oxidation disorder; inborn errors of metabolism; rare disease
MeSH Terms: conditions — Peroxisomal Disorders; Metabolism, Inborn Errors; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
OBJECTIVES:

I. Characterize inheritance patterns of mutations in patients with beta-oxidation disorders.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients undergo clinical and molecular analysis of beta-oxidation enzyme metabolism. The evaluation includes a urinary metabolite profile, and DNA and familial studies.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Beta-oxidation disorder, including: Medium-chain acyl-coenzyme A dehydrogenase deficiency Long-chain 3-hydroxyacyl coenzyme A dehydrogenase deficiency Very-long-chain acyl-coenzyme A dehydrogenase deficiency Short-chain 3-hydroxyacyl coenzyme A dehydrogenase deficiency Long-chain 3-ketoacyl-coenzyme A thiolase deficiency Trifunctional protein deficiency Patient age: 1 day and over

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 1995-09 (Actual); Primary Completion 1998-03-31 (Actual); Study Completion 1998-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold W. Strauss, Study Chair — Washington University School of Medicine

REFERENCES:
- [Background] Wiedermann BL. Acellular pertussis vaccines: what lies ahead? Contemp Pediatr. 1995 Sep;12(9):25-8, 30, 32 passim. PMID 10155576
- [Background] Strauss AW, Jelly DP: The molecular basis of cardiomyopathies due to genetic deficiencies of mitochondrial proteins. pp 323-342.
- [Background] Strauss AW: Defects of mitochondrial proteins and pediatric heart disease. Progress in Pediatric Cardiology 6: 83-90, 1996.
- [Background] Isaacs JD Jr, Sims HF, Powell CK, Bennett MJ, Hale DE, Treem WR, Strauss AW. Maternal acute fatty liver of pregnancy associated with fetal trifunctional protein deficiency: molecular characterization of a novel maternal mutant allele. Pediatr Res. 1996 Sep;40(3):393-8. doi: 10.1203/00006450-199609000-00005. PMID 8865274
- [Background] Strauss AW, Powell CK, Hale DE, Anderson MM, Ahuja A, Brackett JC, Sims HF. Molecular basis of human mitochondrial very-long-chain acyl-CoA dehydrogenase deficiency causing cardiomyopathy and sudden death in childhood. Proc Natl Acad Sci U S A. 1995 Nov 7;92(23):10496-500. doi: 10.1073/pnas.92.23.10496. PMID 7479827
- [Background] Brackett JC, Sims HF, Rinaldo P, Shapiro S, Powell CK, Bennett MJ, Strauss AW. Two alpha subunit donor splice site mutations cause human trifunctional protein deficiency. J Clin Invest. 1995 May;95(5):2076-82. doi: 10.1172/JCI117894. PMID 7738175
- [Background] Payne RM, Johnson MC, Grant JW, Strauss AW. Toward a molecular understanding of congenital heart disease. Circulation. 1995 Jan 15;91(2):494-504. doi: 10.1161/01.cir.91.2.494. PMID 7805255
- [Background] Strauss AW, Johnson MC. The genetic basis of pediatric cardiovascular disease. Semin Perinatol. 1996 Dec;20(6):564-76. doi: 10.1016/s0146-0005(96)80069-3. PMID 9090781
- [Background] Johnson MC, Payne RM, Grant JW, Strauss AW. The genetic basis of paediatric heart disease. Ann Med. 1995 Jun;27(3):289-300. doi: 10.3109/07853899509002580. PMID 7546617
- [Background] Leone TC, Cresci S, Carter ME, Zhang Z, Lala DS, Strauss AW, Kelly DP. The human medium chain Acyl-CoA dehydrogenase gene promoter consists of a complex arrangement of nuclear receptor response elements and Sp1 binding sites. J Biol Chem. 1995 Jul 7;270(27):16308-14. doi: 10.1074/jbc.270.27.16308. PMID 7608198
- [Background] Weinberger MJ, Rinaldo P, Strauss AW, Bennett MJ. Intact alpha-subunit is required for membrane-binding of human mitochondrial trifunctional beta-oxidation protein, but is not necessary for conferring 3-ketoacyl-CoA thiolase activity to the beta-subunit. Biochem Biophys Res Commun. 1995 Apr 6;209(1):47-52. doi: 10.1006/bbrc.1995.1468. PMID 7726862
- [Background] Brackett JC, Sims HF, Steiner RD, Nunge M, Zimmerman EM, deMartinville B, Rinaldo P, Slaugh R, Strauss AW. A novel mutation in medium chain acyl-CoA dehydrogenase causes sudden neonatal death. J Clin Invest. 1994 Oct;94(4):1477-83. doi: 10.1172/JCI117486. PMID 7929823
- [Background] Ziadeh R, Hoffman EP, Finegold DN, Hoop RC, Brackett JC, Strauss AW, Naylor EW. Medium chain acyl-CoA dehydrogenase deficiency in Pennsylvania: neonatal screening shows high incidence and unexpected mutation frequencies. Pediatr Res. 1995 May;37(5):675-8. doi: 10.1203/00006450-199505000-00021. PMID 7603790
- [Background] Peterson KL, Sergienko EE, Wu Y, Kumar NR, Strauss AW, Oleson AE, Muhonen WW, Shabb JB, Srivastava DK. Recombinant human liver medium-chain acyl-CoA dehydrogenase: purification, characterization, and the mechanism of interactions with functionally diverse C8-CoA molecules. Biochemistry. 1995 Nov 14;34(45):14942-53. doi: 10.1021/bi00045a039. PMID 7578106
- [Background] Zhang Z, Zhou Y, Mendelsohn NJ, Bauer GS, Strauss AW. Regulation of the human long chain acyl-CoA dehydrogenase gene by nuclear hormone receptor transcription factors. Biochim Biophys Acta. 1997 Jan 3;1350(1):53-64. doi: 10.1016/s0167-4781(96)00141-8. PMID 9003458
- [Background] Eder M, Krautle F, Dong Y, Vock P, Kieweg V, Kim JJ, Strauss AW, Ghisla S. Characterization of human and pig kidney long-chain-acyl-CoA dehydrogenases and their role in beta-oxidation. Eur J Biochem. 1997 May 1;245(3):600-7. doi: 10.1111/j.1432-1033.1997.00600.x. PMID 9182995
- [Background] Ibdah JA, Tein I, Dionisi-Vici C, Bennett MJ, IJlst L, Gibson B, Wanders RJ, Strauss AW. Mild trifunctional protein deficiency is associated with progressive neuropathy and myopathy and suggests a novel genotype-phenotype correlation. J Clin Invest. 1998 Sep 15;102(6):1193-9. doi: 10.1172/JCI2091. PMID 9739053
- [Background] Kieweg V, Krautle FG, Nandy A, Engst S, Vock P, Abdel-Ghany AG, Bross P, Gregersen N, Rasched I, Strauss A, Ghisla S. Biochemical characterization of purified, human recombinant Lys304-->Glu medium-chain acyl-CoA dehydrogenase containing the common disease-causing mutation and comparison with the normal enzyme. Eur J Biochem. 1997 Jun 1;246(2):548-56. doi: 10.1111/j.1432-1033.1997.00548.x. PMID 9208949
- [Background] Djordjevic S, Dong Y, Paschke R, Frerman FE, Strauss AW, Kim JJ. Identification of the catalytic base in long chain acyl-CoA dehydrogenase. Biochemistry. 1994 Apr 12;33(14):4258-64. doi: 10.1021/bi00180a021. PMID 8155643
- [Background] Kelly DP, Strauss AW. Inherited cardiomyopathies. N Engl J Med. 1994 Mar 31;330(13):913-9. doi: 10.1056/NEJM199403313301308. No abstract available. PMID 8114864